CLINICAL TRIAL: NCT04473352
Title: Diagnostic Accuracy of COVID-19 Detection Tests in Different Body Fluids of Infected Men and Concordance With Viral Cultures
Brief Title: COVID-19 Detection Tests in Different Body Fluids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara (Other)
Collaborators: Universidade Federal do Ceará (Unknown)
Responsible Party: Principal Investigator, Ricardo Reges Maia de Oliveira, PhD, Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara
Other Study IDs: COVID Fluids
Record Dates: First submitted 2020-06-18; First posted 2020-07-16 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: Covid; Body Fluids; Viral Cultures; Detection Tests
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Semen, urine, and saliva: Semen samples will be obtained by the patient through masturbation, and collected in sterile containers. Urine samples will be collected from the medium stream at least 4 hours without emptying the bladder. Saliva samples will be obtained by the swab. The first sample will be collected in the first 14 days after the onset of symptoms and the others on a monthly basis. After 2 consecutive negative samples, no more samples will be taken. Only the virus will be researched using qRT-PCR. Peripheral blood: Samples of peripheral blood are collected through peripheral venipuncture. These samples will be collected at the time of inclusion in the study to assess the viral load, and 45 days after the onset of symptoms to determine the serum levels of sex hormones.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group: Patients with suspected acute viral status for COVID 19 will be invited to participate in the identification of the first symptoms. The diagnosis of COVID-19 will be confirmed according to the determinations of the MS through the reaction of qRT-PCR in the nasopharynx swab. Patients will undergo multiple collections of biological material including blood, saliva, semen, and urine. Each patient will be subjected to serial sample collections. The samples will be processed and analyzed for the presence of viral RNA. Patients with 2 consecutive negative samples did not need to perform subsequent collections.

SUMMARY:
A clinical and experimental study will be carried out in which the clinician will investigate the PCR of the virus early in different body fluids (blood, semen, urine, saliva) and monitor its experimental clearance and evaluate in vitro diagnostic tests and inhibitory factors of viral proliferation.

DETAILED DESCRIPTION:
The World Health Organization (WHO) declared Coronavirus 2019 (COVID-19) as a pandemic on March 11, 2020. Due to the rapid spread of the severe acute respiratory syndrome coronavirus 2 virus (SARS-CoV-2), we are currently facing an unprecedented global situation. One of the main pillars in the control of an epidemic is the performance of large-scale tests providing a quick and accurate diagnosis so that the authorities can take timely action. Therefore, tests for COVID-19 should be prompt, widely available, and implemented outside the hospital environment, to avoid overloading the health system and decreasing the risks of hospital transmission to other patients and health professionals. Although universal testing is a cornerstone for reducing the burden of COVID-19, the accuracy of the commercially available tests for COVID-19 in Brazil remains uncertain. In addition, the natural history of the disease in the different organs and tissues is not unquestionably known, nor because the virus develops better in some tissues and not others. There are still many unanswered questions regarding COVID-19. allow more accurate knowledge of the natural history of the disease in the timeline taking into account the acute and long-term phases. Several families of viruses can affect the male genitourinary system, as is the case of the Zika (ZKV) and Ebola viruses. There are reports that in young patients infected with ZKV, the virus persists in semen for up to 6 months after the symptomatic condition. The other SARS-CoV-1 itself was detected in human testicles associated with an inflammatory process (orchiepididymitis), suggesting the possibility that these viruses could also be detected in the semen. As SARS-CoV-1 was able to overcome the hemato-gestural barrier and induce severe testicular damage in the previous outbreak, it is possible that men infected with COVID-19 may also have testicular damage. Another question that remains unanswered is whether the coronavirus can remain in the body of people considered recovered from Covid-19 for an indefinite period. It is also unknown whether there are molecules in the body fluids capable of inhibiting viral growth. The expected benefits are related to a better understanding of COVID's natural history19 and which body fluids can contribute to understanding the pathophysiology of the disease. It will be possible to identify the best time and the test with the best accuracy to diagnose the disease. It is our intention to identify substances in body fluids with an antiviral effect

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 years
* Agreement with the IC

Exclusion Criteria:

* History of previous prostate surgery or vasectomy
* Inability to assess participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult male patients with suspected acute viral status for COVID 19 of the city of Fortaleza, Ceara, Brazil, who agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Covid19 Detection | September 2021
  Numerical variables will be described by measurements of central tendency (mean or median) and the respective dispersion measurements. Categorical variables will be described by their absolute values, percentages, or proportions. To compare the differences of continuous variables, we will use the Student t-test or the Mann-Whitney test. For comparison of categorical data, we will use the chi-square test. Univariable and multivariable analyses will be performed to identify predictors of COVID-19 detection.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Reges, PhD, Principal Investigator — Nucleo de Pesquisa e Desenvolvimento de Medicamentos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koh D, Cunningham AC. Counting Coronavirus Disease 2019 (COVID-19) Cases: Case Definitions, Screened Populations and Testing Techniques Matter. Ann Acad Med Singap. 2020 Mar;49(3):161-165. PMID 32301478
- [Background] Lin C, Xiang J, Yan M, Li H, Huang S, Shen C. Comparison of throat swabs and sputum specimens for viral nucleic acid detection in 52 cases of novel coronavirus (SARS-Cov-2)-infected pneumonia (COVID-19). Clin Chem Lab Med. 2020 Jun 25;58(7):1089-1094. doi: 10.1515/cclm-2020-0187. PMID 32301745
- [Background] Ling Y, Xu SB, Lin YX, Tian D, Zhu ZQ, Dai FH, Wu F, Song ZG, Huang W, Chen J, Hu BJ, Wang S, Mao EQ, Zhu L, Zhang WH, Lu HZ. Persistence and clearance of viral RNA in 2019 novel coronavirus disease rehabilitation patients. Chin Med J (Engl). 2020 May 5;133(9):1039-1043. doi: 10.1097/CM9.0000000000000774. PMID 32118639
- [Background] Lippi G, Simundic AM, Plebani M. Potential preanalytical and analytical vulnerabilities in the laboratory diagnosis of coronavirus disease 2019 (COVID-19). Clin Chem Lab Med. 2020 Jun 25;58(7):1070-1076. doi: 10.1515/cclm-2020-0285. PMID 32172228
- [Background] Liu R, Ma Q, Han H, Su H, Liu F, Wu K, Wang W, Zhu C. The value of urine biochemical parameters in the prediction of the severity of coronavirus disease 2019. Clin Chem Lab Med. 2020 Jun 25;58(7):1121-1124. doi: 10.1515/cclm-2020-0220. PMID 32286242
- [Background] Mardani R, Ahmadi Vasmehjani A, Zali F, Gholami A, Mousavi Nasab SD, Kaghazian H, Kaviani M, Ahmadi N. Laboratory Parameters in Detection of COVID-19 Patients with Positive RT-PCR; a Diagnostic Accuracy Study. Arch Acad Emerg Med. 2020 Apr 4;8(1):e43. eCollection 2020. PMID 32259132
- [Background] Padoan A, Cosma C, Sciacovelli L, Faggian D, Plebani M. Analytical performances of a chemiluminescence immunoassay for SARS-CoV-2 IgM/IgG and antibody kinetics. Clin Chem Lab Med. 2020 Jun 25;58(7):1081-1088. doi: 10.1515/cclm-2020-0443. PMID 32301749
- [Background] Pan F, Xiao X, Guo J, Song Y, Li H, Patel DP, Spivak AM, Alukal JP, Zhang X, Xiong C, Li PS, Hotaling JM. No evidence of severe acute respiratory syndrome-coronavirus 2 in semen of males recovering from coronavirus disease 2019. Fertil Steril. 2020 Jun;113(6):1135-1139. doi: 10.1016/j.fertnstert.2020.04.024. Epub 2020 Apr 17. PMID 32482249
- [Background] Wang W, Xu Y, Gao R, Lu R, Han K, Wu G, Tan W. Detection of SARS-CoV-2 in Different Types of Clinical Specimens. JAMA. 2020 May 12;323(18):1843-1844. doi: 10.1001/jama.2020.3786. PMID 32159775
- [Background] Wolfel R, Corman VM, Guggemos W, Seilmaier M, Zange S, Muller MA, Niemeyer D, Jones TC, Vollmar P, Rothe C, Hoelscher M, Bleicker T, Brunink S, Schneider J, Ehmann R, Zwirglmaier K, Drosten C, Wendtner C. Virological assessment of hospitalized patients with COVID-2019. Nature. 2020 May;581(7809):465-469. doi: 10.1038/s41586-020-2196-x. Epub 2020 Apr 1. PMID 32235945
- [Background] Wu J, Liu J, Li S, Peng Z, Xiao Z, Wang X, Yan R, Luo J. Detection and analysis of nucleic acid in various biological samples of COVID-19 patients. Travel Med Infect Dis. 2020 Sep-Oct;37:101673. doi: 10.1016/j.tmaid.2020.101673. Epub 2020 Apr 18. PMID 32311437
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Yu F, Yan L, Wang N, Yang S, Wang L, Tang Y, Gao G, Wang S, Ma C, Xie R, Wang F, Tan C, Zhu L, Guo Y, Zhang F. Quantitative Detection and Viral Load Analysis of SARS-CoV-2 in Infected Patients. Clin Infect Dis. 2020 Jul 28;71(15):793-798. doi: 10.1093/cid/ciaa345. PMID 32221523
- [Result] Castro R, Luz PM, Wakimoto MD, Veloso VG, Grinsztejn B, Perazzo H. COVID-19: a meta-analysis of diagnostic test accuracy of commercial assays registered in Brazil. Braz J Infect Dis. 2020 Mar-Apr;24(2):180-187. doi: 10.1016/j.bjid.2020.04.003. Epub 2020 Apr 18. PMID 32330437
- [Result] Chen Y, Chen L, Deng Q, Zhang G, Wu K, Ni L, Yang Y, Liu B, Wang W, Wei C, Yang J, Ye G, Cheng Z. The presence of SARS-CoV-2 RNA in the feces of COVID-19 patients. J Med Virol. 2020 Jul;92(7):833-840. doi: 10.1002/jmv.25825. Epub 2020 Apr 25. PMID 32243607
- [Result] Infantino M, Grossi V, Lari B, Bambi R, Perri A, Manneschi M, Terenzi G, Liotti I, Ciotta G, Taddei C, Benucci M, Casprini P, Veneziani F, Fabbri S, Pompetti A, Manfredi M. Diagnostic accuracy of an automated chemiluminescent immunoassay for anti-SARS-CoV-2 IgM and IgG antibodies: an Italian experience. J Med Virol. 2020 Sep;92(9):1671-1675. doi: 10.1002/jmv.25932. Epub 2020 May 10. PMID 32330291